CLINICAL TRIAL: NCT06361563
Title: Patients With Upper Gastrointestinal Cancer Enrolled in a Patient Support Program to Receive Nivolumab in the Adjuvant Setting: Real World Data From Canada
Brief Title: Real-World Use of Adjuvant Nivolumab in Patients With Upper Gastrointestinal Cancer in Canada
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-1442
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Upper Gastrointestinal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants treated with adjuvant nivolumab
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — As per product label

SUMMARY:
The purpose of this observational study is to describe the patient, disease and treatment characteristics of eligible participants with upper gastrointestinal cancer treated with adjuvant nivolumab.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in Bristol-Myers Squibb GastroEsophageal Opdivo in Resected Patients with Residual Pathological Disease Patient Support Program (GEORge PSP) in Canada
* Patients who have consented to the use of their de-identified data generated from information collected in the course of the GEORge PSP

Exclusion Criteria:

* Aged <18 years
* Did not receive concurrent chemoradiotherapy prior to surgery
* Positive margins following resection
* No residual disease following complete resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is comprised of individuals diagnosed with Stage II or III esophageal cancer (EC) or gastroesophageal junction cancer (GEJC) that participated in the Bristol-Myers Squibb Patient Support Program (PSP) in Canada, GEORge PSP (GastroEsophageal Opdivo in Resected patients with residual pathological disease).
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Participant sociodemographics | Baseline
Participant Eastern Cooperative Oncology Group (ECOG) score | Baseline
Participant histology results | Baseline
Participant comorbidities | Baseline
Participant tumour location | Baseline
Date of tumour resection | Baseline
Participant primary upper gastrointestinal cancer diagnosis | Baseline

SECONDARY OUTCOMES:
Initial nivolumab dosage prescribed to participants | Index date
Number of nivolumab treatments received | Up to 484 days
Nivolumab dosage modification | Up to 484 days
Nivolumab treatment duration | Up to 484 days
Reason for participant discharge | Up to 484 days
Participant adverse events (AEs) | Up to 484 days
Management of participant adverse events (AEs) | Up to 484 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Bayshore Specialty Rx Ltd., Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts